CLINICAL TRIAL: NCT04742556
Title: A Phase I Open-label Trial of BI 3011441 in Japanese Patients With NRAS/KRAS Mutation Positive Advanced, Unresectable or Metastatic Refractory Solid Tumours
Brief Title: A Study to Test Different Doses of BI 3011441 in Japanese People With Different Types of Advanced Cancer (NRAS/KRAS Mutation Positive)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1469-0002
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumors, KRAS Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 mg BI 3011441 (Experimental): The patients were administered 4 milligram (mg) BI 3011441 soft capsule once daily during 4 weeks with water limited to a maximum of 100 milliliters (mL) per capsules, taken without food, at least 1 hour before a meal or 1 hour after a meal. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: BI 3011441
- 6 mg BI 3011441 (Experimental): The patients were administered 6 milligram (mg) BI 3011441 soft capsule once daily during 4 weeks with water limited to a maximum of 100 milliliters (mL) per capsules, taken without food, at least 1 hour before a meal or 1 hour after a meal. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: BI 3011441
- 8 mg BI 3011441 (Experimental): The patients were administered 8 milligram (mg) BI 3011441 soft capsule once daily during 4 weeks with water limited to a maximum of 100 milliliters (mL) per capsules, taken without food, at least 1 hour before a meal or 1 hour after a meal. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: BI 3011441

INTERVENTIONS:
Drug: BI 3011441 — BI 3011441

SUMMARY:
This study is open to Japanese adults with different types of advanced cancer that are positive for NRAS/KRAS mutations. This is a study in people for whom previous treatment was not successful or no standard treatment exists.

The purpose of this study is to find the highest dose of BI 3011441 that Japanese people with advanced cancer can tolerate. BI 3011441 is a medicine that may turn off a signal by NRAS/KRAS that makes tumours grow.

Participants take BI 3011441 as capsules once a day. Participants can stay in the study as long as they benefit from treatment and can tolerate it. The doctors collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 20 years of age at screening.
* Signed and dated written informed consent in accordance with Good Clinical Practice(GCP) and local legislation prior to admission to the trial.
* Pathologically documented, locally-advanced or metastatic malignancy with previously identified activating Neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS) or Kirsten rat sarcoma viral oncogene homologue (KRAS) mutation based on local test.
* Provision of archival tumor tissue, if available, to confirm retrospectively NRAS or KRAS mutation status and for biomarker assessment.
* Willingness to undergo pre- and on-treatment tumour biopsies for pharmacodynamics and biomarker assessment. Patients can be enrolled without tumour biopsy upon agreement between the Investigator and the Sponsor if tumour biopsy is not feasible (Apply only to study site which agreed to conduct biopsy).
* Must have either progressed despite appropriate prior standard therapies or for whom no standard therapy exists for their tumour type and disease stage
* Must have at least one target lesion that can be measured per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Further inclusion criteria apply.

Exclusion Criteria:

* Previous anticancer chemotherapy within 3 weeks of the first administration of trial drug. Previous anticancer hormonal treatment or anticancer immunotherapy within 2 weeks of the first administration of trial drugs.
* Radiotherapy within 4 weeks prior to first administration of BI 3011441 except as follows

  * Palliative radiotherapy to regions other than the chest is allowed up to 2 weeks prior to start of treatment
  * Single dose palliative radiotherapy for symptomatic metastasis within 2 weeks prior to start of treatment may be allowed but must be discussed with the sponsor.
* Major surgery within 4 weeks prior to start of treatment or scheduled during the projected course of the trial
* Previous treatment with a Rat sarcoma (RAS), Mitogen-activated protein kinase (MAPK) targeting agent
* Previous treatment with any investigational agent(s) or targeted treatment within 4 weeks (28 days) prior to start of trial drug or concurrent participation in another clinical trial with an investigational device or drug.
* Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the study medications
* Patients who have a history or current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment or central serous retinopathy; for example, predisposing factors of RVO or central serous retinopathy include uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes.
* Patients who have visible retinal pathology that is considered a risk factor for RVO or central serous retinopathy as assessed by ophthalmic examination, such as:

  * Evidence of new optic disc cupping
  * Evidence of new visual field defects
  * Intraocular pressure >21 mm Hg History or presence of cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of ≥2, unstable angina or poorly controlled arrhythmia which are considered as clinically relevant by the investigator; Myocardial infarction within 6 months prior to start of treatment. Uncontrolled hypertension is defined as: Blood pressure (BP) measured in a rested and relaxed condition, where systolic BP >=140 mmHg, or diastolic BP >= 90 mmHg, with or without medication.

Further exclusion criteria apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a phase 1, open-label trial of BI 3011441 monotherapy dose escalation of Maximum tolerated dose (MTD) determination in Japanese patients with Neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS)/Kirsten rat sarcoma viral oncogene homologue (KRAS) mutation positive advanced for whom previous treatment was not successful or no standard treatment exists, unresectable or metastatic refractory solid tumours.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441 | 8 mg BI 3011441
Started | 3 | 4 | 8
Completed | 0 | 0 | 0
Not Completed | 3 | 4 | 8
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Clinical disease progression | 0 | 1 | 2
Not completed — Objective disease progression | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This set included all patients who were dispensed trial medication (BI 3011441) and were documented to have taken at least 1 dose of open-label trial medication (BI 3011441).
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441 | 8 mg BI 3011441 | Total
Number analyzed (Participants) | 3 | 4 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (13.9) | 55.5 (13.3) | 49.5 (13.8) | 53.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 6
  Male | 2 | 3 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With DLTs in the MTD Evaluation Period
Description: Number of participants with Dose limiting toxicities (DLT) occurring during the first treatment cycle (first 4 weeks). DLT was defined as any of the following adverse events related to the treatment:
  * Haematologic toxicities:
  * Neutropenia Grade 4 lasting for >7 days days without documented infection
  * Neutropenia Grade ≥3 with documented infection
  * Grade ≥3 febrile neutropenia
  * Grade 4 neutropenia defined as life-threatening consequences or urgent intervention indicated
  * Grade 5 neutropenia defined as a fatal neutropenia
  * Grade 3 thrombocytopenia associated with bleeding
Time Frame: First treatment cycle, the first 28 days following the start of trial medication.
Population: Maximum tolerated dose (MTD) evaluation set: Included all patients from the treated set who were not replaced and were evaluable for the MTD evaluation. Only patients with evaluable DLTs are reported.
Measure: Count of Participants; unit: Participants
Groups:
- 6 mg BI 3011441Edit: The patients were administered 6 milligram (mg) BI 3011441 soft capsule once daily during 4 weeks with water limited to a maximum of 100 milliliters (mL) per capsules, taken without food, at least 1 hour before a meal or 1 hour after a meal. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 2
Statistical Analysis 1: Comparison: 4 mg BI 3011441; Probability of true DLT rate was determined using a Bayesian 2-parameter logistic regression model with overdose control; Test type: Other; Probability of true DLT rate in [0.33-1] = 0.0051
Statistical Analysis 2: Comparison: 6 mg BI 3011441Edit; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of true DLT rate in [0.33-1] = 0.03105
Statistical Analysis 3: Comparison: 8 mg BI 3011441; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of true DLT rate in [0.33-1] = 0.27405

2. Primary Outcome: Maximum Tolerated Dose (MTD) of BI 3011441 Monotherapy
Description: Maximum tolerated dose (MTD) of BI 3011441 monotherapy. The MTD was defined as the highest dose with less than 25% risk of the true dose-limiting toxicity (DLT) rate being equal or above 0.33 (EWOC criterion) during the MTD evaluation period. The analysis of the MTD was based on a Bayesian 2-parameter logistic regression model (BLRM) with overdose control.
Time Frame: First treatment cycle, the first 28 days following the start of trial medication.
Population: Maximum tolerated dose (MTD) evaluation set: Included all patients from the treated set who were not replaced and were evaluable for the MTD evaluation. Only evaluable for DLTs patients were considered in the analysis.
Measure: Number; unit: milligram (mg)
Groups:
- BI 3011441: This arm comprises all participants in this trial who were administered 4, 6, 8 mg BI 3011441. The patients were administered BI 3011441 soft capsule once daily during 4 weeks with water limited to a maximum of 100 milliliters (mL) per capsules, taken without food, at least 1 hour before a meal or 1 hour after a meal. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
Arm/Group | BI 3011441
Number analyzed (Participants) | 12
milligram (mg) | NA — Maximum tolerated dose was not reached during the MTD evaluation period (the first 28 days of study treatment).

3. Secondary Outcome: Number of Patients With DLTs During the Entire On-treatment Period
Description: as for outcome 1
Time Frame: From first BI 3011441 intake until last BI 3011441 intake + 30 days of Residual effect period (REP), up to 373 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 3 | 4 | 8
Participants | 0 | 0 | 2

4. Secondary Outcome: Number of Patients With Grade ≥3 Treatment-related Adverse Events
Description: Number of participants with Grade ≥3 treatment-related adverse events is reported. The severity of AEs were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. The CTCAE grades are Grade 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first BI 3011441 intake until last BI 3011441 intake + 30 days of Residual effect period (REP), up to 373 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441 | 8 mg BI 3011441
Number analyzed (Participants) | 3 | 4 | 8
Participants
  Grade 3 | 1 | 4 | 6
  Grade 4 | 0 | 0 | 1
  Grade 5 | 1 | 0 | 0

5. Secondary Outcome: Number of Patients With Treatment Related Adverse Events
Description: Number of participants with drug-related adverse events (AEs) analysed as investigator defined drug-related AEs is presented. Medical judgment was used to determine the relationship between the AEs and the study medication, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.
Time Frame: From first BI 3011441 intake until last BI 3011441 intake + 30 days of Residual effect period (REP), up to 373 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 3 | 4 | 8
Participants | 3 | 3 | 8

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 3011441 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 3011441 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: Cycle 1: Day 1: Within 5 minutes (min) before and 30min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h and optionally 12h. and Day 2 : Within 5 minutes (min) before dosing on Day 2.
Population: Pharmacokinetic parameter analysis set (PKS): Includes all subjects in the treated set who provided at least one evaluable observation for at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomol/ milliliter (h*nmol/mL)
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 3 | 4 | 8
hour * nanomol/ milliliter (h*nmol/mL) | 246 (28.2) | 471 (35.3) | 704 (39.6)

7. Secondary Outcome: Area Under the Concentration-time Curve of BI 3011441 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point at Steady State (AUC0-tz,ss)
Description: Area under the concentration-time curve of BI 3011441 in plasma over the time interval from 0 to the last quantifiable data point at steady state (AUC0-tz,ss) is reported.
Time Frame: Cycle 1: Day 15: Within 5 minutes (min) before drug administration on Day 15, and 30min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h and optionally 12h. and Day 16 : Within 5 minutes (min) before dosing on Day 16.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomol/ milliliter (h*nmol/mL)
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 2 | 3 | 4
hour * nanomol/ milliliter (h*nmol/mL) | 505 (8.89) | 973 (22.9) | 833 (54.7)

8. Secondary Outcome: Maximum Measured Concentration of BI 3011441 in Plasma After First Dose (Cmax)
Description: Maximum measured concentration of BI 3011441 in plasma (Cmax) is reported.
Time Frame: as for outcome 6
Population: Pharmacokinetic parameter analysis set (PKS): Includes all subjects in the treated set who provided at least one evaluable observation for at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/ liter (nmol/L)
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 3 | 4 | 8
nanomol/ liter (nmol/L) | 72.3 (11.8) | 91.8 (27.1) | 133 (32.6)

9. Secondary Outcome: Maximum Measured Concentration of BI 3011441 in Plasma at Steady State (Cmax,ss)
Description: Maximum measured concentration of BI 3011441 in plasma at steady state (Cmax,ss) is reported. PK samples were collected at the following timepoints.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/ liter (nmol/L)
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441Edit | 8 mg BI 3011441
Number analyzed (Participants) | 2 | 3 | 4
nanomol/ liter (nmol/L) | 73.5 (12.1) | 124 (37.2) | 130 (54.9)

ADVERSE EVENTS:
Time Frame: From first BI 3011441 intake until last BI 3011441 intake + 30 days of Residual effect period (REP), up to 373 days.
Description: Treated Set (TS): This set included all patients who were dispensed trial medication (BI 3011441) and were documented to have taken at least 1 dose of open-label trial medication (BI 3011441).
Arm/Group | 4 mg BI 3011441 | 6 mg BI 3011441 | 8 mg BI 3011441
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/4 | 6/8
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg BI 3011441 (N=3) | 6 mg BI 3011441 (N=4) | 8 mg BI 3011441 (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Serous retinal detachment (Eye disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg BI 3011441 (N=3) | 6 mg BI 3011441 (N=4) | 8 mg BI 3011441 (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 4
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 2
Malaise (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04742556/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04742556/SAP_001.pdf